CLINICAL TRIAL: NCT05301049
Title: Prevalence, Severity, Risk Factors, and Prognostic Value of Hyponatremia in Patients With Traumatic Brain Injury : a Retrospective Cohort Study.
Brief Title: Prevalence, Severity, Risk Factors, and Prognostic Value of Hyponatremia in Patients With Traumatic Brain Injury
Acronym: WATERWAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0011
Record Dates: First submitted 2022-02-07; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Traumatic Brain Injury
Keywords: Hyponatremia; Syndrome of Inappropriate Anti Diuretic Hormone (SIADH); Cerebral Salt Waste Syndrome (CSW)
MeSH Terms: conditions — Brain Injuries, Traumatic; Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hyponatremia (HN) is the most common electrolytic disorder in the traumatic brain injury (TBI) population, found in 17 to 51% of patients according to the series. Two etiologies predominate in the literature, the Syndrome of Inappropriate Anti Diuretic Hormone (SIADH) and the Cerebral Salt Waste Syndrome (CSW), but none has been precisely described in terms of epidemiology, risk factors or severity. Moreover, SIADH and CSH were often confused in previous works.

The main goal of our study is to assess retrospectively prevalence, severity, time to onset, length, risk factors of HN in a large population of TBI patients, as well as treatment modalities and prognosis. A specific distinction was performed between SIADH or CSW.

DETAILED DESCRIPTION:
This is a retrospective descriptive study.

The included patients will be those admitted in the trauma intensive care unit of Lapeyronie University Hospital (Montpellier, France) with a TBI (head AIS ≥1) during a period of 4 years, 01/01/2014 to 31/12/2017.

Using our databank the investigators estimate 650 to 700 patients who met inclusion criteria during this period and will be analyzed. Inclusions will be confirmed after the opening of medical records.

Definition of SIADH is defined as the occurrence of a hyponatremia (≤135 mmol/L) associated with inappropriate urine concentration (urinary/plasmatic osmolarity ≥1) and a low daily urine volume (<1500 ml/24H).

Definition of CSW is defined as the occurrence of a hyponatremia (≤135 mmol/L) associated with a massive natriuresis (>140 mmol/L) and a daily urine volume > 1500 ml/24H.

Data collection will concern the medical records: medical history, traumatism severity, cerebral injuries on computed tomography, severe complications, specific treatments, and biological course from ICU admission to discharge.

The main endpoint will be the prevalence of hyponatremia (≤135 mmol/L) in the first 10 days after the traumatic brain injury.

The secondary endpoints will be the prevalence specific prevalence of CSW and SIADH, risk factors of these nosological entities, their severity, their timing to onset and their morbimorality.

ELIGIBILITY:
Inclusion criteria:

* âge ≥ 18 years
* presence of traumatic brain injury at the ICU admission

Exclusion criteria:

* Discharged from ICU or death < 48 hours from the admission
* Lack of data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in the trauma intensive care unit of the Lapeyronie university hospital (Montpellier, France) with a traumatic brain injury Period of 4 years between 01/01/2014 and 31/12/2017.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-28 (Estimated); Study Completion 2022-07-28 (Estimated)

PRIMARY OUTCOMES:
Occurrence of hyponatremia | during the 10 first days after the traumatic brain injury
  Hyponatremia ≤ 135mmol/L

SECONDARY OUTCOMES:
Occurrence SIADH | during the 10 first days after the traumatic brain injury
  Hyponatremia ≤ 135mmol/L associated with inappropriate urine concentration (urinary/plasmatic osmolarity ≥1) and a low daily urine volume (<1500 ml/24H).
Occurrence CSW | during the 10 first days after the traumatic brain injury
  Hyponatremia (≤135 mmol/L) associated with a massive natriuresis (>140 mmol/L) and a daily urine volume > 1500 ml/24H
Determination of risk factors of hyponatremia | during the 10 first days after the traumatic brain injury
  Traumatics injuries, early management, early complications, sodium and water intakes, treatments.
Morbi-mortality | Day 1 (Hospitalization)
  Death, duration of mechanical ventilation, duration of renal replacement therapy, length of ICU stay and length of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan CHARBIT, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, Montepllier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC